CLINICAL TRIAL: NCT05942677
Title: Comparison of Flat Colorectal Lesion Detection by Artificial Intelligence-assisted Colonoscopy Versus Endoscopists: AIChallenge - Medtronic
Brief Title: Comparison of Flat Colorectal Lesion Detection by Artificial Intelligence-assisted Colonoscopy Versus Endoscopists
Acronym: AIChallengeMed
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_1366
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Flat Colorectal Lesion
Keywords: detection; AI; CAD; colorectal cancer; LST; adenoma; SSL
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Colorectal lesion diagnostic: Every patient referred to our center for colorectal endoscopy for investigation and/or resection of colorectal lesion can join the cohort of this study and will benefit from diagnosis and treatment by experienced endoscopists.
  Interventions: Procedure: proportion of colorectal lesions

INTERVENTIONS:
Procedure: proportion of colorectal lesions — Evaluation of the proportion of colorectal lesions detected by a computer-aided detection system (CADe) compared with experienced endoscopists.

SUMMARY:
The development of artificial intelligence (AI) systems in the field of colorectal endoscopy is currently booming, colorectal cancer being, by its frequency and severity, a real public health problem.

In terms of image analysis, AI is indeed able to perform many tasks simultaneously (lesion detection, classification, and segmentation) and to combine them.

Lesion detection is thus the starting point of the whole chain to choose at the end the most appropriate treatment for the patient. Large-scale studies have demonstrated the superiority of artificial intelligence-assisted detection over the usual detection by gastroenterologists, mainly for the detection of sub-centimeter polyps.

However, the investigators have shown that a recent computer-aided detection system (CADe) such as the ENDO-AID software in combination with the EVIS X1 video column (Olympus, Tokyo, Japan) may present difficulties in the detection of flat lesions such as sessile serrated lesions (SSLs) and non-granular laterally spreading tumors (LST-NGs).

This represents a major challenge because in addition to their shape being difficult to identify for the human eye in practice and where AI assistance would be of great value, these rare lesions are associated with advanced histology.

In addition, the investigators recently described the case of a worrisome false negative of AI-assisted colonoscopy, which failed to detect a flat adenocarcinoma in the transverse colon.

Therefore, it is important to measure the false negative rate of AI detection based on the macroscopic shape of the lesion. Comparing this rate to the human endoscopist's false negatives would improve the performance of AI for this specific lesion subtype in the future.

ELIGIBILITY:
Inclusion Criteria:

* both gender patients even or older than 18 years old
* patient with French Health Insurance coverage
* obtaining of oral non opposition to research after loyal, clear and complete delivery of information
* patients addressed to our center for colorectal lesion resection
* patients presenting a colorectal lesion discovered during a diagnostic colonoscopy

Exclusion Criteria:

* patients with health disorders needing short procedure times
* patients with no colorectal lesion
* difficulty continuing colonoscopy due to poor sedation
* difficulty continuing colonoscopy due to a serious adverse event
* inappropriate participation after colonoscopy is completed
* unwillingness to participate after colonoscopy is completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Every patient referred to our center for colorectal endoscopy for investigation and/or resection of colorectal lesion can join the cohort of this study and will benefit from diagnosis and treatment by experienced endoscopists.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the proportion of colorectal lesions | Time point can be reached either 2 weeks after endoscopic resection or between 2-4 months later in case of surgery
  Evaluation of the proportion of colorectal lesions detected by a computer-aided detection system (CADe) compared with experienced endoscopists and correlation with final histology reading.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Edouard Herriot, Lyon, France